CLINICAL TRIAL: NCT05059171
Title: Postoperative Pain After Pulpectomy of Primary Molars Using With Rotary Versus Reciprocation Motions of Two Single Files: A Randomized Clinical Trial
Brief Title: Postoperative Pain of Rotary Versus Reciprocating Motions of Two Single Files
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahmad Elheeny, Associate Professor, Minia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 122/2020
Record Dates: First submitted 2021-09-13; First posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rotary motion using OneShape single file (Active Comparator): File size 25 with a taper of 0.06 was mounted to a 6:1 speed-reduction headpiece powered by X Smart Plus endomotor (Dentsply Maillefer, Ballaigues, Switzerland). The speed and torque were set to 400 rpm and 1 N.cm torque, respectively. In a picking motion without pressure, mechanical preparation began with the first RC two-thirds followed by the next 3 mm followed by the full WL.
  Interventions: Device: OneSahpe single file
- Reciprocating motion using WaveOne Gold single file (Active Comparator): A Primary file size 25 a taper of 0.07 was installed to pre-programmed reciprocation angles and speed for the WaveOne system handpiece of an endomotor (X Smart Plus endomotor (Dentsply Maillefer, Ballaigues, Switzerland). After ensuring a passive fit of the hand file along the predetermined WL, the RC coronal two-thirds was initially instrumented then followed by the full WL.
  Interventions: Device: WaveOne Gold single file

INTERVENTIONS:
Device: OneSahpe single file — The rotary motion of OneShape single file
  Arms: Rotary motion using OneShape single file
Device: WaveOne Gold single file — reciprocation motions of WaveOne Gold single file
  Arms: Reciprocating motion using WaveOne Gold single file

SUMMARY:
An equivalent parallel randomized clinical trial was approved by the local University Committee of Ethics. 260 children with necrotic primary molars were allocated into 2 equal groups (82 children per group). The participants were allocated into two groups; group "1" teeth were instrumented with OneShape rotary system (Micro Mega, Besancon, France), and group "2" teeth were instrumented with WaveOne Gold reciprocating system (Dentsply Maillefer, Ballaigues, Switzerland). Postoperative pain was assessed using a four-point pain intensity rating scale adopted from Wong-Baker FACES (WBF) pain scale . The face scale consists of four faces with a brief title describing each face representing a scale from the first face (score 1), second face (score 2), third face (score 3), and forth face (score 4) 3. Postoperative pain was assessed at 6 six time intervals (at 6, 12, 24, 48, 72 hours and one-week).

ELIGIBILITY:
Inclusion Criteria:

1. Children ages from 4 to 8 years classified as class I or II according to the American Society of Anesthesiologists (ASA).
2. No previous dental experience.
3. Non-vital primary molar (necrotic or with chronic apical periodontitis) which confirmed radiographicly with the presence or absence of periapical radiolucency.
4. Severe tooth mobility.

Exclusion Criteria:

1. Severe behaviour or emotional disabilities.
2. Analgesic intake in the preceding 12 hours.
3. Non-restorable crowns of primary molars.
4. Radiographic presence of internal root resorption or massive bone destruction.
5. Root resorption exceeded one-third of the root length.

   -

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — children aged from 4 to 8 years
Enrollment: 260 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | One week
  Postoperative pain was assessed using a four-point pain intensity rating scale adopted from Wong-Baker FACES (WBF) pain scale . The face scale consists of four faces with a brief title describing each face representing a scale from the first face (score 1), second face (score 2), third face (score 3), and fourth face (score 4) 17. Postoperative pain was assessed at 6 six time intervals

CONTACTS AND LOCATIONS:
Locations (1):
- Ngwa Khattab, Minya, Minya Governorate, Egypt